CLINICAL TRIAL: NCT04663555
Title: Effect of Dexamethasone in Patients With ARDS and COVID-19 - Prospective, Multi-centre, Open-label, Parallel-group, Randomized Controlled Trial (REMED Trial)
Brief Title: Effect of Two Different Doses of Dexamethasone in Patients With ARDS and COVID-19
Acronym: REMED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other); Vascular surgery, University hospital Královské Vinohrady, Prague (Other); General University Hospital, Prague (Other); University Hospital Ostrava (Other); St. Anne's University Hospital Brno (Unknown); Motol University Hospital (Other); University Hospital Olomouc (Other); University Hospital Plzeň (Unknown); Tomáš Baťa Regional Hospital (Unknown); Military University Hospital Praha (Unknown)
Responsible Party: Principal Investigator, Jan Malaska, MD. Ph.D. EDIC, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZECRIN No. 2020/47; 2020-005887-70 (EudraCT Number)
Record Dates: First submitted 2020-12-09; First posted 2020-12-11 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Covid19; ARDS
Keywords: Covid19; ARDS; dexamethasone
MeSH Terms: conditions — COVID-19 | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: REMED is a prospective phase II open-label randomized controlled trial testing superiority of dexamethasone 20 mg vs 6 mg. The study is multi-centre and will be conducted in intensive care units (ICUs) of university hospitals in the Czech Republic. The trial aims to be pragmatic, i.e. designed to evaluate the effectiveness of the intervention in conditions that are very close to the real-life routine clinical practice. Dexamethasone will be administered once daily intravenously for 10 days. 300 participants will be enrolled and followed up for 360 days after randomization.
  Following stratification factors will be applied:
  * Age < 65 and ≥ 65 (12);
  * Charlson Comorbidity index (CCI; APPENDIX B Assessment tools, scores, and scales, Chapter 14.2) < 3 and ≥ 3;
  * CRP < 150 mg/L and ≥ 150 mg/L
  * Trial centre. Patients will be randomized in 1 : 1 ratio in one of the two treatment arms. Randomization through eCRF will be available 24 hours every day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEX 20 mg (Experimental): Patients in the intervention group after randomization will receive dexamethasone 20 mg intravenously once daily on day 1-5, followed by dexamethasone 10 mg intravenously once daily on day 6-10.
  Interventions: Drug: Dexamethasone
- DEX 6 mg (Active Comparator): Patients in the control group after randomization will receive dexamethasone 6 mg day 1-10.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Patients in the intervention group after randomization will receive dexamethasone 20 mg intravenously once daily on day 1-5, followed by dexamethasone 10 mg intravenously once daily on day 6-10. If successful extubation occurs before day 10, treatment with dexamethasone is withdrawn.

SUMMARY:
REMED is a prospective, phase II, open-label, randomised controlled trial testing superiority of dexamethasone 20 mg vs 6 mg. The trial aims to be pragmatic, i.e. designed to evaluate the effectiveness of the intervention in conditions that are close to real-life routine clinical practice. The study is multi-centre and will be conducted in the intensive care units (ICUs) of ten university hospitals in the Czech Republic. This is an open-label trial in which the participants and the study staff will be aware of the allocated intervention. Blinded pre-planned statistical analysis will be performed.

DETAILED DESCRIPTION:
Since December 2019, Covid-19 virus has infected millions of people worldwide. A significant number of patients develop hyperinflammatory state affecting lungs, which may lead to the need of oxygen therapy. In most severe cases, acute respiratory distress syndrome (ARDS) develops and high flow oxygen therapy or invasive mechanical ventilation is necessary (Wu et al., 2020). Therapeutic options in Covid-19 associated ARDS patients remain limited and mortality is still excessive. Systemic corticosteroids have potential to limit hyperinflammatory response by modulating immune system. This effect is mediated mainly by binding to glucocorticosteroid receptor α (GRα)(Meduri et al., 2020). Their effectiveness was proved in heterogeneous ARDS patients recently (Villar et al., 2020). In patients with Covid-19 pneumonia in need for oxygen therapy or mechanical ventilation, dexamethasone 6 mg per day is currently recommended. This therapy is mandated by the results of RECOVERY trial (Horby et al., 2020). After this trial was published, three randomised trials comparing hydrocortisone (Angus et al., 2020; Dequin et al., 2020) or dexamethasone (Tomazini et al., 2020) against placebo were stopped prematurely. All these studies were included in the subsequent IPD metaanalysis (Sterne et al., 2020). However, dose of 6 mg of dexamethasone is currently being reappraised. The aforementioned study in non Covid-19 ARDS patients (Villar et al., 2020) used 20 mg of dexamethasone per day, which is roughly equivalent to the methylprednisolone regimen (1mg/kg/day) studied in early severe ARDS patients (Meduri et al., 2007). Only these moderate doses (80-100 mg of methylprednisolone, equivalent to 15-19 mg of dexamethasone) have full potential to modulate immune response by saturating GRα receptors (Meduri et al., 2020). Importantly, prematurely stopped CoDEX trial (Tomazini et al., 2020) comparing dexamethasone against placebo in Covid-ARDS patients, used initial daily dose of 20 mg of dexamethasone versus placebo.

In the light of these facts, 6 mg of dexamethasone given to COVID-19 patients with different severity of illness (WHO classification group 5-10) may miss important therapeutic potential or may prevent a potential deleterious effects of a full dose therapeutic corticosteroid. Authors hypothesize that the patients with moderate to severe ARDS undergoing mechanical ventilation may benefit from higher doses of dexamethasone (Villar et al., 2020; Tomazini et al., 2020; Meduri et al., 2007).

The primary objective of this study is to test the hypothesis that administration of dexamethasone 20 mg is superior over 6 mg in adult patients with moderate or severe ARDS due to confirmed COVID-19.

Primary endpoint: Number of ventilator-free days (VFDs) at 28 days after randomisation, defined as being alive and free from mechanical ventilation (more than 48 hours).

Secondary endpoints:

1. Mortality from any cause at 60 days after randomization;
2. Dynamics of inflammatory marker (CRP) change from Day 1 to Day 14;
3. WHO Clinical Progression Scale at Day 14 (range 0-10; 0 = no illness, 1-9 = increasing level of care, and 10 = death);
4. Adverse events related to corticosteroids (new infections, new thrombotic complications) until Day 28 or hospital discharge;
5. Independence at 90 days after randomization assessed by Barthel Index The long-term outcomes of this study are to assess long-term consequences on mortality and quality of life at 180 and 360 days through telephone structured interview using Barthel Index.

ELIGIBILITY:
Inclusion criteria:

Subjects will be eligible for the trial if they meet all of the following criteria:

1. Adult (≥ 18 years of age) at time of enrolment;
2. Present COVID-19 (infection confirmed by RT-PCR or antigen testing);
3. Intubation/mechanical ventilation or ongoing high-flow nasal cannula (HFNC) oxygen therapy;
4. Moderate or severe ARDS according to Berlin criteria:

   * Moderate - PaO2/FiO2 100-200 mmHg;
   * Severe - PaO2/FiO2 < 100 mmHg;
5. Admission to ICU in the last 24 hours.

Exclusion criteria:

Subjects will not be eligible for the trial if they meet any of the following criteria:

1. Known allergy/hypersensitivity to dexamethasone or excipients of the investigational medicinal product (e.g. parabens, benzyl alcohol);
2. Fulfilled criteria for ARDS for ≥ 14 days at enrolment;
3. Pregnancy or breastfeeding;
4. Unwillingness to comply with contraception measurements from the enrolment to at least 1 week after the last dose of dexamethasone (sexual abstinence is considered as the adequate contraception method);
5. End-of-life decision or patient is expected to die within next 24 hours;
6. Decision not to intubate or ceilings of treatment in place;
7. Immunosuppression and/or immunosuppressive drugs in medical history:

   1. Systemic immunosuppressive drugs or chemotherapy in the past 30 days;
   2. Systemic corticosteroids use before hospitalization;
   3. Any dose of dexamethasone during the present hospital stay for COVID-19 for more than (≥) last 5 days before enrolment;
   4. Systemic corticosteroids during present hospital stay for other conditions than COVID-19 (e.g. septic shock);
8. Present haematological or generalized solid malignancy;
9. Any of contraindications of corticosteroids, e.g.

   * intractable hyperglycaemia;
   * active gastrointestinal bleeding;
   * adrenal gland disorders;
   * a presence of superinfection diagnosed with locally established clinical and laboratory criteria without adequate antimicrobial treatment;
10. Cardiac arrest before ICU admission;
11. Participation in another interventional trial in the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Number of ventilator-free days (VFDs) at 28 days after randomization | 28 days
  Number of ventilator-free days (VFDs) at 28 days after randomisation, defined as being alive and free from mechanical ventilation (more than 48 hours)

SECONDARY OUTCOMES:
Mortality from any cause at 60 days after randomization | 60 days
WHO clinical progression scale at day 14 | 14 days
  WHO clinical progression scale (range, 0-10, where 0 = no illness, 1-9 = increasing level of care, and 10 = death) (WHO Working Group on the Clinical Characterisation and Management of COVID-19 infection, 2020) assessed at day 14
Dynamics of inflammatory marker | 14 days
  Dynamics of inflammatory marker (CRP) change from Day 1 to Day 14
Adverse events related to corticosteroids | 28 days
  new infections, new thrombotic complications
Functional independence | 90 days
  Independence at 90 days after randomization assessed by Barthel Index

OTHER OUTCOMES:
Long-term outcome regarding mortality | 180 and 360 days
  Death from any cause at 180 and 360 days
Long-term outcome regarding functional independence | 180 and 360 days
  Functional independence at 180 and 360 days assesed through telephone structured interview using Barthel Index.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Collected data will be shared with other ongoing clinical trials on the same topic for individual patient ́s data (IPD) metaanalysis or shared upon relevant requests. Also de-identified participant-level dataset will be made available 6 months after the publication of the results of the study at www.mendeley.com
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: De-identified participant-level dataset will be made available 6 months after the publication of the results of the study at www.mendeley.com
Access Criteria: Planned IPD metaanalysis or other relevant request

REFERENCES:
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Meduri GU, Annane D, Confalonieri M, Chrousos GP, Rochwerg B, Busby A, Ruaro B, Meibohm B. Pharmacological principles guiding prolonged glucocorticoid treatment in ARDS. Intensive Care Med. 2020 Dec;46(12):2284-2296. doi: 10.1007/s00134-020-06289-8. Epub 2020 Nov 4. PMID 33150472
- [Background] Villar J, Ferrando C, Martinez D, Ambros A, Munoz T, Soler JA, Aguilar G, Alba F, Gonzalez-Higueras E, Conesa LA, Martin-Rodriguez C, Diaz-Dominguez FJ, Serna-Grande P, Rivas R, Ferreres J, Belda J, Capilla L, Tallet A, Anon JM, Fernandez RL, Gonzalez-Martin JM; dexamethasone in ARDS network. Dexamethasone treatment for the acute respiratory distress syndrome: a multicentre, randomised controlled trial. Lancet Respir Med. 2020 Mar;8(3):267-276. doi: 10.1016/S2213-2600(19)30417-5. Epub 2020 Feb 7. PMID 32043986
- [Background] RECOVERY Collaborative Group; Horby P, Lim WS, Emberson JR, Mafham M, Bell JL, Linsell L, Staplin N, Brightling C, Ustianowski A, Elmahi E, Prudon B, Green C, Felton T, Chadwick D, Rege K, Fegan C, Chappell LC, Faust SN, Jaki T, Jeffery K, Montgomery A, Rowan K, Juszczak E, Baillie JK, Haynes R, Landray MJ. Dexamethasone in Hospitalized Patients with Covid-19. N Engl J Med. 2021 Feb 25;384(8):693-704. doi: 10.1056/NEJMoa2021436. Epub 2020 Jul 17. PMID 32678530
- [Background] Angus DC, Derde L, Al-Beidh F, Annane D, Arabi Y, Beane A, van Bentum-Puijk W, Berry L, Bhimani Z, Bonten M, Bradbury C, Brunkhorst F, Buxton M, Buzgau A, Cheng AC, de Jong M, Detry M, Estcourt L, Fitzgerald M, Goossens H, Green C, Haniffa R, Higgins AM, Horvat C, Hullegie SJ, Kruger P, Lamontagne F, Lawler PR, Linstrum K, Litton E, Lorenzi E, Marshall J, McAuley D, McGlothin A, McGuinness S, McVerry B, Montgomery S, Mouncey P, Murthy S, Nichol A, Parke R, Parker J, Rowan K, Sanil A, Santos M, Saunders C, Seymour C, Turner A, van de Veerdonk F, Venkatesh B, Zarychanski R, Berry S, Lewis RJ, McArthur C, Webb SA, Gordon AC; Writing Committee for the REMAP-CAP Investigators; Al-Beidh F, Angus D, Annane D, Arabi Y, van Bentum-Puijk W, Berry S, Beane A, Bhimani Z, Bonten M, Bradbury C, Brunkhorst F, Buxton M, Cheng A, De Jong M, Derde L, Estcourt L, Goossens H, Gordon A, Green C, Haniffa R, Lamontagne F, Lawler P, Litton E, Marshall J, McArthur C, McAuley D, McGuinness S, McVerry B, Montgomery S, Mouncey P, Murthy S, Nichol A, Parke R, Rowan K, Seymour C, Turner A, van de Veerdonk F, Webb S, Zarychanski R, Campbell L, Forbes A, Gattas D, Heritier S, Higgins L, Kruger P, Peake S, Presneill J, Seppelt I, Trapani T, Young P, Bagshaw S, Daneman N, Ferguson N, Misak C, Santos M, Hullegie S, Pletz M, Rohde G, Rowan K, Alexander B, Basile K, Girard T, Horvat C, Huang D, Linstrum K, Vates J, Beasley R, Fowler R, McGloughlin S, Morpeth S, Paterson D, Venkatesh B, Uyeki T, Baillie K, Duffy E, Fowler R, Hills T, Orr K, Patanwala A, Tong S, Netea M, Bihari S, Carrier M, Fergusson D, Goligher E, Haidar G, Hunt B, Kumar A, Laffan M, Lawless P, Lother S, McCallum P, Middeldopr S, McQuilten Z, Neal M, Pasi J, Schutgens R, Stanworth S, Turgeon A, Weissman A, Adhikari N, Anstey M, Brant E, de Man A, Lamonagne F, Masse MH, Udy A, Arnold D, Begin P, Charlewood R, Chasse M, Coyne M, Cooper J, Daly J, Gosbell I, Harvala-Simmonds H, Hills T, MacLennan S, Menon D, McDyer J, Pridee N, Roberts D, Shankar-Hari M, Thomas H, Tinmouth A, Triulzi D, Walsh T, Wood E, Calfee C, O'Kane C, Shyamsundar M, Sinha P, Thompson T, Young I, Bihari S, Hodgson C, Laffey J, McAuley D, Orford N, Neto A, Detry M, Fitzgerald M, Lewis R, McGlothlin A, Sanil A, Saunders C, Berry L, Lorenzi E, Miller E, Singh V, Zammit C, van Bentum Puijk W, Bouwman W, Mangindaan Y, Parker L, Peters S, Rietveld I, Raymakers K, Ganpat R, Brillinger N, Markgraf R, Ainscough K, Brickell K, Anjum A, Lane JB, Richards-Belle A, Saull M, Wiley D, Bion J, Connor J, Gates S, Manax V, van der Poll T, Reynolds J, van Beurden M, Effelaar E, Schotsman J, Boyd C, Harland C, Shearer A, Wren J, Clermont G, Garrard W, Kalchthaler K, King A, Ricketts D, Malakoutis S, Marroquin O, Music E, Quinn K, Cate H, Pearson K, Collins J, Hanson J, Williams P, Jackson S, Asghar A, Dyas S, Sutu M, Murphy S, Williamson D, Mguni N, Potter A, Porter D, Goodwin J, Rook C, Harrison S, Williams H, Campbell H, Lomme K, Williamson J, Sheffield J, van't Hoff W, McCracken P, Young M, Board J, Mart E, Knott C, Smith J, Boschert C, Affleck J, Ramanan M, D'Souza R, Pateman K, Shakih A, Cheung W, Kol M, Wong H, Shah A, Wagh A, Simpson J, Duke G, Chan P, Cartner B, Hunter S, Laver R, Shrestha T, Regli A, Pellicano A, McCullough J, Tallott M, Kumar N, Panwar R, Brinkerhoff G, Koppen C, Cazzola F, Brain M, Mineall S, Fischer R, Biradar V, Soar N, White H, Estensen K, Morrison L, Smith J, Cooper M, Health M, Shehabi Y, Al-Bassam W, Hulley A, Whitehead C, Lowrey J, Gresha R, Walsham J, Meyer J, Harward M, Venz E, Williams P, Kurenda C, Smith K, Smith M, Garcia R, Barge D, Byrne D, Byrne K, Driscoll A, Fortune L, Janin P, Yarad E, Hammond N, Bass F, Ashelford A, Waterson S, Wedd S, McNamara R, Buhr H, Coles J, Schweikert S, Wibrow B, Rauniyar R, Myers E, Fysh E, Dawda A, Mevavala B, Litton E, Ferrier J, Nair P, Buscher H, Reynolds C, Santamaria J, Barbazza L, Homes J, Smith R, Murray L, Brailsford J, Forbes L, Maguire T, Mariappa V, Smith J, Simpson S, Maiden M, Bone A, Horton M, Salerno T, Sterba M, Geng W, Depuydt P, De Waele J, De Bus L, Fierens J, Bracke S, Reeve B, Dechert W, Chasse M, Carrier FM, Boumahni D, Benettaib F, Ghamraoui A, Bellemare D, Cloutier E, Francoeur C, Lamontagne F, D'Aragon F, Carbonneau E, Leblond J, Vazquez-Grande G, Marten N, Wilson M, Albert M, Serri K, Cavayas A, Duplaix M, Williams V, Rochwerg B, Karachi T, Oczkowski S, Centofanti J, Millen T, Duan E, Tsang J, Patterson L, English S, Watpool I, Porteous R, Miezitis S, McIntyre L, Brochard L, Burns K, Sandhu G, Khalid I, Binnie A, Powell E, McMillan A, Luk T, Aref N, Andric Z, Cviljevic S, Dimoti R, Zapalac M, Mirkovic G, Barsic B, Kutlesa M, Kotarski V, Vujaklija Brajkovic A, Babel J, Sever H, Dragija L, Kusan I, Vaara S, Pettila L, Heinonen J, Kuitunen A, Karlsson S, Vahtera A, Kiiski H, Ristimaki S, Azaiz A, Charron C, Godement M, Geri G, Vieillard-Baron A, Pourcine F, Monchi M, Luis D, Mercier R, Sagnier A, Verrier N, Caplin C, Siami S, Aparicio C, Vautier S, Jeblaoui A, Fartoukh M, Courtin L, Labbe V, Leparco C, Muller G, Nay MA, Kamel T, Benzekri D, Jacquier S, Mercier E, Chartier D, Salmon C, Dequin P, Schneider F, Morel G, L'Hotellier S, Badie J, Berdaguer FD, Malfroy S, Mezher C, Bourgoin C, Megarbane B, Voicu S, Deye N, Malissin I, Sutterlin L, Guitton C, Darreau C, Landais M, Chudeau N, Robert A, Moine P, Heming N, Maxime V, Bossard I, Nicholier TB, Colin G, Zinzoni V, Maquigneau N, Finn A, Kress G, Hoff U, Friedrich Hinrichs C, Nee J, Pletz M, Hagel S, Ankert J, Kolanos S, Bloos F, Petros S, Pasieka B, Kunz K, Appelt P, Schutze B, Kluge S, Nierhaus A, Jarczak D, Roedl K, Weismann D, Frey A, Klinikum Neukolln V, Reill L, Distler M, Maselli A, Belteczki J, Magyar I, Fazekas A, Kovacs S, Szoke V, Szigligeti G, Leszkoven J, Collins D, Breen P, Frohlich S, Whelan R, McNicholas B, Scully M, Casey S, Kernan M, Doran P, O'Dywer M, Smyth M, Hayes L, Hoiting O, Peters M, Rengers E, Evers M, Prinssen A, Bosch Ziekenhuis J, Simons K, Rozendaal W, Polderman F, de Jager P, Moviat M, Paling A, Salet A, Rademaker E, Peters AL, de Jonge E, Wigbers J, Guilder E, Butler M, Cowdrey KA, Newby L, Chen Y, Simmonds C, McConnochie R, Ritzema Carter J, Henderson S, Van Der Heyden K, Mehrtens J, Williams T, Kazemi A, Song R, Lai V, Girijadevi D, Everitt R, Russell R, Hacking D, Buehner U, Williams E, Browne T, Grimwade K, Goodson J, Keet O, Callender O, Martynoga R, Trask K, Butler A, Schischka L, Young C, Lesona E, Olatunji S, Robertson Y, Jose N, Amaro dos Santos Catorze T, de Lima Pereira TNA, Neves Pessoa LM, Castro Ferreira RM, Pereira Sousa Bastos JM, Aysel Florescu S, Stanciu D, Zaharia MF, Kosa AG, Codreanu D, Marabi Y, Al Qasim E, Moneer Hagazy M, Al Swaidan L, Arishi H, Munoz-Bermudez R, Marin-Corral J, Salazar Degracia A, Parrilla Gomez F, Mateo Lopez MI, Rodriguez Fernandez J, Carcel Fernandez S, Carmona Flores R, Leon Lopez R, de la Fuente Martos C, Allan A, Polgarova P, Farahi N, McWilliam S, Hawcutt D, Rad L, O'Malley L, Whitbread J, Kelsall O, Wild L, Thrush J, Wood H, Austin K, Donnelly A, Kelly M, O'Kane S, McClintock D, Warnock M, Johnston P, Gallagher LJ, Mc Goldrick C, Mc Master M, Strzelecka A, Jha R, Kalogirou M, Ellis C, Krishnamurthy V, Deelchand V, Silversides J, McGuigan P, Ward K, O'Neill A, Finn S, Phillips B, Mullan D, Oritz-Ruiz de Gordoa L, Thomas M, Sweet K, Grimmer L, Johnson R, Pinnell J, Robinson M, Gledhill L, Wood T, Morgan M, Cole J, Hill H, Davies M, Antcliffe D, Templeton M, Rojo R, Coghlan P, Smee J, Mackay E, Cort J, Whileman A, Spencer T, Spittle N, Kasipandian V, Patel A, Allibone S, Genetu RM, Ramali M, Ghosh A, Bamford P, London E, Cawley K, Faulkner M, Jeffrey H, Smith T, Brewer C, Gregory J, Limb J, Cowton A, O'Brien J, Nikitas N, Wells C, Lankester L, Pulletz M, Williams P, Birch J, Wiseman S, Horton S, Alegria A, Turki S, Elsefi T, Crisp N, Allen L, McCullagh I, Robinson P, Hays C, Babio-Galan M, Stevenson H, Khare D, Pinder M, Selvamoni S, Gopinath A, Pugh R, Menzies D, Mackay C, Allan E, Davies G, Puxty K, McCue C, Cathcart S, Hickey N, Ireland J, Yusuff H, Isgro G, Brightling C, Bourne M, Craner M, Watters M, Prout R, Davies L, Pegler S, Kyeremeh L, Arbane G, Wilson K, Gomm L, Francia F, Brett S, Sousa Arias S, Elin Hall R, Budd J, Small C, Birch J, Collins E, Henning J, Bonner S, Hugill K, Cirstea E, Wilkinson D, Karlikowski M, Sutherland H, Wilhelmsen E, Woods J, North J, Sundaran D, Hollos L, Coburn S, Walsh J, Turns M, Hopkins P, Smith J, Noble H, Depante MT, Clarey E, Laha S, Verlander M, Williams A, Huckle A, Hall A, Cooke J, Gardiner-Hill C, Maloney C, Qureshi H, Flint N, Nicholson S, Southin S, Nicholson A, Borgatta B, Turner-Bone I, Reddy A, Wilding L, Chamara Warnapura L, Agno Sathianathan R, Golden D, Hart C, Jones J, Bannard-Smith J, Henry J, Birchall K, Pomeroy F, Quayle R, Makowski A, Misztal B, Ahmed I, KyereDiabour T, Naiker K, Stewart R, Mwaura E, Mew L, Wren L, Willams F, Innes R, Doble P, Hutter J, Shovelton C, Plumb B, Szakmany T, Hamlyn V, Hawkins N, Lewis S, Dell A, Gopal S, Ganguly S, Smallwood A, Harris N, Metherell S, Lazaro JM, Newman T, Fletcher S, Nortje J, Fottrell-Gould D, Randell G, Zaman M, Elmahi E, Jones A, Hall K, Mills G, Ryalls K, Bowler H, Sall J, Bourne R, Borrill Z, Duncan T, Lamb T, Shaw J, Fox C, Moreno Cuesta J, Xavier K, Purohit D, Elhassan M, Bakthavatsalam D, Rowland M, Hutton P, Bashyal A, Davidson N, Hird C, Chhablani M, Phalod G, Kirkby A, Archer S, Netherton K, Reschreiter H, Camsooksai J, Patch S, Jenkins S, Pogson D, Rose S, Daly Z, Brimfield L, Claridge H, Parekh D, Bergin C, Bates M, Dasgin J, McGhee C, Sim M, Hay SK, Henderson S, Phull MK, Zaidi A, Pogreban T, Rosaroso LP, Harvey D, Lowe B, Meredith M, Ryan L, Hormis A, Walker R, Collier D, Kimpton S, Oakley S, Rooney K, Rodden N, Hughes E, Thomson N, McGlynn D, Walden A, Jacques N, Coles H, Tilney E, Vowell E, Schuster-Bruce M, Pitts S, Miln R, Purandare L, Vamplew L, Spivey M, Bean S, Burt K, Moore L, Day C, Gibson C, Gordon E, Zitter L, Keenan S, Baker E, Cherian S, Cutler S, Roynon-Reed A, Harrington K, Raithatha A, Bauchmuller K, Ahmad N, Grecu I, Trodd D, Martin J, Wrey Brown C, Arias AM, Craven T, Hope D, Singleton J, Clark S, Rae N, Welters I, Hamilton DO, Williams K, Waugh V, Shaw D, Puthucheary Z, Martin T, Santos F, Uddin R, Somerville A, Tatham KC, Jhanji S, Black E, Dela Rosa A, Howle R, Tully R, Drummond A, Dearden J, Philbin J, Munt S, Vuylsteke A, Chan C, Victor S, Matsa R, Gellamucho M, Creagh-Brown B, Tooley J, Montague L, De Beaux F, Bullman L, Kersiake I, Demetriou C, Mitchard S, Ramos L, White K, Donnison P, Johns M, Casey R, Mattocks L, Salisbury S, Dark P, Claxton A, McLachlan D, Slevin K, Lee S, Hulme J, Joseph S, Kinney F, Senya HJ, Oborska A, Kayani A, Hadebe B, Orath Prabakaran R, Nichols L, Thomas M, Worner R, Faulkner B, Gendall E, Hayes K, Hamilton-Davies C, Chan C, Mfuko C, Abbass H, Mandadapu V, Leaver S, Forton D, Patel K, Paramasivam E, Powell M, Gould R, Wilby E, Howcroft C, Banach D, Fernandez de Pinedo Artaraz Z, Cabreros L, White I, Croft M, Holland N, Pereira R, Zaki A, Johnson D, Jackson M, Garrard H, Juhaz V, Roy A, Rostron A, Woods L, Cornell S, Pillai S, Harford R, Rees T, Ivatt H, Sundara Raman A, Davey M, Lee K, Barber R, Chablani M, Brohi F, Jagannathan V, Clark M, Purvis S, Wetherill B, Dushianthan A, Cusack R, de Courcy-Golder K, Smith S, Jackson S, Attwood B, Parsons P, Page V, Zhao XB, Oza D, Rhodes J, Anderson T, Morris S, Xia Le Tai C, Thomas A, Keen A, Digby S, Cowley N, Wild L, Southern D, Reddy H, Campbell A, Watkins C, Smuts S, Touma O, Barnes N, Alexander P, Felton T, Ferguson S, Sellers K, Bradley-Potts J, Yates D, Birkinshaw I, Kell K, Marshall N, Carr-Knott L, Summers C. Effect of Hydrocortisone on Mortality and Organ Support in Patients With Severe COVID-19: The REMAP-CAP COVID-19 Corticosteroid Domain Randomized Clinical Trial. JAMA. 2020 Oct 6;324(13):1317-1329. doi: 10.1001/jama.2020.17022. PMID 32876697
- [Background] Dequin PF, Heming N, Meziani F, Plantefeve G, Voiriot G, Badie J, Francois B, Aubron C, Ricard JD, Ehrmann S, Jouan Y, Guillon A, Leclerc M, Coffre C, Bourgoin H, Lengelle C, Caille-Fenerol C, Tavernier E, Zohar S, Giraudeau B, Annane D, Le Gouge A; CAPE COVID Trial Group and the CRICS-TriGGERSep Network. Effect of Hydrocortisone on 21-Day Mortality or Respiratory Support Among Critically Ill Patients With COVID-19: A Randomized Clinical Trial. JAMA. 2020 Oct 6;324(13):1298-1306. doi: 10.1001/jama.2020.16761. PMID 32876689
- [Background] Tomazini BM, Maia IS, Cavalcanti AB, Berwanger O, Rosa RG, Veiga VC, Avezum A, Lopes RD, Bueno FR, Silva MVAO, Baldassare FP, Costa ELV, Moura RAB, Honorato MO, Costa AN, Damiani LP, Lisboa T, Kawano-Dourado L, Zampieri FG, Olivato GB, Righy C, Amendola CP, Roepke RML, Freitas DHM, Forte DN, Freitas FGR, Fernandes CCF, Melro LMG, Junior GFS, Morais DC, Zung S, Machado FR, Azevedo LCP; COALITION COVID-19 Brazil III Investigators. Effect of Dexamethasone on Days Alive and Ventilator-Free in Patients With Moderate or Severe Acute Respiratory Distress Syndrome and COVID-19: The CoDEX Randomized Clinical Trial. JAMA. 2020 Oct 6;324(13):1307-1316. doi: 10.1001/jama.2020.17021. PMID 32876695
- [Background] WHO Rapid Evidence Appraisal for COVID-19 Therapies (REACT) Working Group; Sterne JAC, Murthy S, Diaz JV, Slutsky AS, Villar J, Angus DC, Annane D, Azevedo LCP, Berwanger O, Cavalcanti AB, Dequin PF, Du B, Emberson J, Fisher D, Giraudeau B, Gordon AC, Granholm A, Green C, Haynes R, Heming N, Higgins JPT, Horby P, Juni P, Landray MJ, Le Gouge A, Leclerc M, Lim WS, Machado FR, McArthur C, Meziani F, Moller MH, Perner A, Petersen MW, Savovic J, Tomazini B, Veiga VC, Webb S, Marshall JC. Association Between Administration of Systemic Corticosteroids and Mortality Among Critically Ill Patients With COVID-19: A Meta-analysis. JAMA. 2020 Oct 6;324(13):1330-1341. doi: 10.1001/jama.2020.17023. PMID 32876694
- [Background] Meduri GU, Golden E, Freire AX, Taylor E, Zaman M, Carson SJ, Gibson M, Umberger R. Methylprednisolone infusion in early severe ARDS: results of a randomized controlled trial. Chest. 2007 Apr;131(4):954-63. doi: 10.1378/chest.06-2100. PMID 17426195
- [Background] Harhay MO, Casey JD, Clement M, Collins SP, Gayat E, Gong MN, Jaber S, Laterre PF, Marshall JC, Matthay MA, Monroe RE, Rice TW, Rubin E, Self WH, Mebazaa A. Contemporary strategies to improve clinical trial design for critical care research: insights from the First Critical Care Clinical Trialists Workshop. Intensive Care Med. 2020 May;46(5):930-942. doi: 10.1007/s00134-020-05934-6. Epub 2020 Feb 18. PMID 32072303
- [Background] Yehya N, Harhay MO, Curley MAQ, Schoenfeld DA, Reeder RW. Reappraisal of Ventilator-Free Days in Critical Care Research. Am J Respir Crit Care Med. 2019 Oct 1;200(7):828-836. doi: 10.1164/rccm.201810-2050CP. PMID 31034248
- [Background] WHO Working Group on the Clinical Characterisation and Management of COVID-19 infection. A minimal common outcome measure set for COVID-19 clinical research. Lancet Infect Dis. 2020 Aug;20(8):e192-e197. doi: 10.1016/S1473-3099(20)30483-7. Epub 2020 Jun 12. PMID 32539990
- [Derived] Malaska J, Stasek J, Maca J, Kutej M, Duska F, Kafka P, Klementova O, Doubravska L, Hruda J, Fencl M, Gabrhelik T, Ciz L, Zatloukal J, Pouska J, Novotny P, Balik M, Demlova R, Kubatova J, Vinklerova J, Grodova K, Stepanova R, Svobodnik A, Kratochvil M, Klucka J, Stourac P, Singer M; REMED Study Group. Effects of two different dexamethasone dosing regimens on ventilator-free days and long-term mortality in COVID-19 patients with moderate-to-severe ARDS: the REMED randomized clinical trial. Eur J Med Res. 2024 Dec 23;29(1):616. doi: 10.1186/s40001-024-02215-6. PMID 39710693
- [Derived] Malaska J, Stasek J, Duska F, Balik M, Maca J, Hruda J, Vymazal T, Klementova O, Zatloukal J, Gabrhelik T, Novotny P, Demlova R, Kubatova J, Vinklerova J, Svobodnik A, Kratochvil M, Klucka J, Gal R, Singer M; REMED Study Group. Effect of dexamethasone in patients with ARDS and COVID-19 (REMED trial)-study protocol for a prospective, multi-centre, open-label, parallel-group, randomized controlled trial. Trials. 2022 Jan 15;23(1):35. doi: 10.1186/s13063-021-05963-6. PMID 35033182
- [Derived] Malaska J, Stasek J, Duska F, Balik M, Maca J, Hruda J, Vymazal T, Klementova O, Zatloukal J, Gabrhelik T, Novotny P, Demlova R, Kubatova J, Vinklerova J, Svobodnik A, Kratochvil M, Klucka J, Gal R, Singer M; REMED Study Group. Effect of dexamethasone in patients with ARDS and COVID-19 - prospective, multi-centre, open-label, parallel-group, randomised controlled trial (REMED trial): A structured summary of a study protocol for a randomised controlled trial. Trials. 2021 Mar 1;22(1):172. doi: 10.1186/s13063-021-05116-9. PMID 33648568

DOCUMENTS (1):
  • Study Protocol (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT04663555/Prot_000.pdf